CLINICAL TRIAL: NCT00391898
Title: A 3-month, Multi-center, Double-blind, Randomized Study to Evaluate the Efficacy of Levodopa/Carbidopa/Entacapone vs Levodopa/Carbidopa in Parkinson's Disease Patients With Impairment of Activities of Daily Living and Early Wearing-off With Levodopa
Brief Title: Efficacy of Levodopa/Carbidopa/Entacapone vs Levodopa/Carbidopa in Parkinson's Disease Patients With Early Wearing-off
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CELC200AES03
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Results first posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease, adults, levodopa/carbidopa/entacapone, wearing-off, activities of daily living
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Levodopa/carbidopa/entacapone (Experimental)
  Interventions: Drug: Levodopa/carbidopa/entacapone
- Levodopa/carbidopa (Active Comparator)
  Interventions: Drug: Levodopa/carbidopa

INTERVENTIONS:
Drug: Levodopa/carbidopa/entacapone — Patients were instructed to take the study medication at the same hours and the same levodopa dose they were taking prior to enrollment in this study. Levodopa/carbidopa/entacapone was available in 2 oral dosage forms: 100/25/200 or 150/37.5/200 mg encapsulated tablets.
  Arms: Levodopa/carbidopa/entacapone
Drug: Levodopa/carbidopa — Patients were instructed to take the study medication at the same hours and the same levodopa dose they were taking prior to enrollment in this study. Levodopa/carbidopa was available in 2 oral dosage forms: One or one and one-half 100/25 mg encapsulated tablets.
  Arms: Levodopa/carbidopa

SUMMARY:
The study evaluated the efficacy of levodopa/carbidopa/entacapone vs levodopa/carbidopa in patients with Parkinson's disease and early wearing-off with levodopa

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ages ≥ 30 and ≤ 80 years old.
2. A clinical diagnosis of idiopathic Parkinson's disease.
3. Taking a stable dose of levodopa/carbidopa (≥ 300 and ≤ 600mg) for a period of at least 1 month prior to study entry.
4. Must be using any of the following levodopa/carbidopa standard formulation levodopa/carbidopa 100/25mg dose in any intake of the day.

   * 1 full tablet, and/or
   * 1½ tablets The patient can also be using, for a period of at least 1 month prior to study entry, 1 tablet of the controlled release formulation of levodopa/carbidopa 100/25 mg (marketed in Spain as Sinemet Plus retard) or 1 tablet the controlled release formulation of levodopa/carbidopa 200/50 mg (marketed in Spain as Sinemet retard) in each intake, at different doses.
5. Must have early end-of-dose wearing-off defined by >= 2 or <=7 positive responses to the QUICK questionnaire.
6. Must have a minimum UPDRS part II (ADL) score of 9.
7. Patients without dyskinesia or with mild dyskinesia.
8. Female patients must be either post-menopausal or using one or more acceptable methods of contraception.
9. Must be capable of satisfying the requirements of the protocol and must be willing and able to give informed consent according to legal requirements.

Exclusion Criteria:

1. Previous or current use of entacapone.
2. History, signs, or symptoms suggesting the diagnosis of secondary or atypical parkinsonism.
3. Unstable Parkinson's disease patients.
4. Patients who experience severe dyskinesia.
5. The following levodopa/carbidopa doses and strengths are not permitted:

   * Patients taking ½ tablet of standard formulation levodopa/carbidopa 100/25
   * Patients taking standard formulation levodopa/carbidopa 100/10 or 250/25
   * Patients taking fewer than 3 or more than 6 daily intakes of standard formulation levodopa/carbidopa 100/25 (fewer than 300mg or more than 600mg of levodopa)
6. Patients with hallucinations or psychiatric diseases related to levodopa or dopamine agonists intake. Patients with major depression.
7. Female patients who are pregnant, trying to become pregnant or nursing (lactating) an infant.
8. Concomitant treatment with MAO-inhibitors (except selegiline up to 10mg/day), rotigotine or neuroleptics, within 60 days prior to the screening visit.
9. Patients with a previous history of Neuroleptic Malignant Syndrome (NMS) and/or non-traumatic rhabdomyolysis.
10. Participated in another trial of an investigational drug/device within the last 30 days prior to study entry.
11. Patients who have a history of poor compliance or are in the Investigator's judgment unlikely to comply with medical regimens or study requirements.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Tolosa-Sarró, Dr., Principal Investigator — Hospital Clínic i Provincial de Barcelona
Locations (26):
- Spain (26):
  - Hospital Juan Canalejo, A Coruña
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Fundación Hospital de Alcorcón, Alcorcón (Madrid
  - Hospital General de Alicante, Alicante
  - Centro Médico Teknon, Barcelona
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Corporació Sanitària Parc Taulí Sabadell, Barcelona
  - Hospital General Yagüe, Burgos
  - Policlínica Gipuzkoa, Donostia / San Sebastian
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitari Bellvitge Princeps d'Espanya, L'Hospitalet de Llobregat , Barcelona
  - Clínica Ruber, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Universitaria de Navarra, Pamplona
  - Hospital General de Catalunya, Sant Cugat Del Valles, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario de la Fe, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Gral. de Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levodopa/Carbidopa/Entacapone | Levodopa/Carbidopa
Started | 46 (Safety population for Levodopa/carbidopa/entacapone is 45, for Levodopa/carbidopa, per randomized.) | 49
Completed | 35 | 39
Not Completed | 11 | 10
Not completed — Adverse Event | 3 | 0
Not completed — Other | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levodopa/Carbidopa/Entacapone | Levodopa/Carbidopa | Total
Number analyzed (Participants) | 45 | 49 | 94
Age Continuous [Mean (Standard Deviation); unit: Years] | 66.40 (8.18) | 66.45 (9.04) | 66.43 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline Measure based on Safety population
  Participants
    Female | 25 | 22 | 47
    Male | 20 | 27 | 47
Region of Enrollment [Number; unit: participants] — Baseline measure based on safety population.
  participants
    Spain | 45 | 49 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change in the Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activities of Daily Living [ADL]) Score From Baseline to Month 3
Description: The UPDRS is a standardized assessment scale used to measure a patient's disease state. It is completed by a blinded rater. There are 6 parts to the UPDRS. Part II (items 5-17; total score 0-52, calculated as the sum of the individual items) measures the patient's activities of daily living. A lower total score indicates greater symptom control. A negative change score indicates improvement.
Time Frame: Baseline to end of study (Month 3)
Population: Per Protocol set with the last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Levodopa/Carbidopa/Entacapone | Levodopa/Carbidopa
Number analyzed (Participants) | 35 | 36
Units on a scale | -2.5 (2.8) | -0.5 (3.0)

2. Secondary Outcome: Change in the UPDRS Part I (Mentation, Behavior, and Mood) Score From Baseline to Month 3
Description: The UPDRS is a standardized assessment scale used to measure a patient's disease state. It is completed by a blinded rater. There are 6 parts to the UPDRS. Part I (items 1-4; total score 0-16, calculated as the sum of the individual items) measures the patient's mentation, mood and behavior. A lower total score indicates greater symptom control. A negative change score indicates improvement.
Time Frame: Baseline to end of study (Month 3)
Population: Per Protocol set with LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Levodopa/Carbidopa/Entacapone | Levodopa/Carbidopa
Number analyzed (Participants) | 35 | 36
Units on a scale | -0.5 (1.6) | -0.2 (1.0)

3. Secondary Outcome: Change in the UPDRS Part III (Motor Function) Score From Baseline to Month 3
Description: The UPDRS is a standardized assessment scale used to measure a patient's disease state. It is completed by a blinded rater. There are 6 parts to the UPDRS. Part III (items 18-31; total score 0-56, calculated as the sum of the individual items) measures the patient's motor function. A lower total score indicates greater symptom control. A negative change score indicates improvement.
Time Frame: Baseline to end of study (Month 3)
Population: Per Protocol set with LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Levodopa/Carbidopa/Entacapone | Levodopa/Carbidopa
Number analyzed (Participants) | 35 | 36
Units on a scale | -4.0 (4.6) | -1.42 (5.5)

4. Secondary Outcome: Change in the UPDRS Part IV (Complications of Therapy) Score From Baseline to Month 3
Description: Part IV of the UPDRS measures complications the patient may be experiencing with therapy and was only collected at and after the visit at which the first dyskinesia or episode of wearing-off was recorded. Part IV is composed of 3 sections and 11 items: A (32-35, dyskinesia), B (36-39, clinical fluctuations, C (40-42, other complications) (total score 0-23, calculated as the sum of the individual items). A lower total score indicates greater symptom control. A negative change score indicates improvement.
Time Frame: Baseline to end of study (Month 3)
Population: Per Protocol set with LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Levodopa/Carbidopa/Entacapone | Levodopa/Carbidopa
Number analyzed (Participants) | 35 | 36
Units on a scale | -0.6 (1.8) | -0.1 (1.3)

5. Secondary Outcome: Change in the 39-item Parkinson's Disease Questionnaire (PDQ-39) Total Score From Baseline to Month 3
Description: The PDQ-39 is an instrument used to assess quality of life in individuals with Parkinson's disease. The questionnaire provides scores on eight scales: Mobility, activities of daily living, emotions, stigma, social support, cognitions, communication, and bodily discomfort. Questions are scored on a 5-point Likert scale ranging from 1 (never) to 3 (sometimes) to 5 (always). The total score can range from 39 to 195. A lower score indicates better quality of life. A positive change score indicates an improvement.
Time Frame: Baseline to end of study (Month 3)
Population: Per Protocol set with LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Levodopa/Carbidopa/Entacapone | Levodopa/Carbidopa
Number analyzed (Participants) | 35 | 36
Units on a scale | 6.3 (20.4) | 0.8 (15.6)

6. Secondary Outcome: Patient and Investigator Global Evaluation of the Patient
Description: Both the patient and the investigator made an evaluation of the change in the patient's condition by rating the condition of the patient at the end of the study compared to patient's condition at baseline. The rating was made on a scale ranging from -3 to +3: (-3: Very much improved, -2: much improved, -1: mild improvement, 0: no change, +1: mild deterioration, +2: much deterioration, +3: very much deterioration). A negative score indicates improvement.
Time Frame: Baseline to end of study (Month 3)
Population: Per Protocol set with LOCF
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Levodopa/Carbidopa/Entacapone | Levodopa/Carbidopa
Number analyzed (Participants) | 34 | 35
Units on a scale
  Patient global evaluation | -0.9 (1.1) [-2.0 to 2.0] | -0.4 (1.2) [-2.0 to 2.0]
  Investigator global evaluation | -0.9 (1.0) | -0.3 (0.9)

7. Secondary Outcome: Change on the QUICK Questionnaire (QQ) Score From Baseline to Month 3
Description: The QQ is a self-administered questionnaire that includes 19 wearing-off (WO) symptoms (motor and non-motor). A positive answer to each of the 19 symptoms is given by patients if they presented with a symptom and the symptom disappeared after the next drug dose. Two positive answers are diagnostic of wearing-off (WO). A negative change score indicates improvement.
Time Frame: Baseline to end of study (Month 3)
Population: Per Protocol set with LOCF
Measure: Mean (Standard Deviation); unit: Positive answers
Arm/Group | Levodopa/Carbidopa/Entacapone | Levodopa/Carbidopa
Number analyzed (Participants) | 35 | 36
Positive answers | -0.6 (1.8) | -0.6 (2.3)

ADVERSE EVENTS:
Arm/Group | Levodopa/Carbidopa/Entacapone | Levodopa/Carbidopa
Serious Adverse Events (participants affected / at risk) | 1/45 | 1/49
Other Adverse Events (participants affected / at risk) | 10/45 | 3/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levodopa/Carbidopa/Entacapone (N=45) | Levodopa/Carbidopa (N=49)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Delusion (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levodopa/Carbidopa/Entacapone (N=45) | Levodopa/Carbidopa (N=49)
Retching (Gastrointestinal disorders) | 3 | 2
Dyskinesia (Nervous system disorders) | 7 | 1
Anxiety (Psychiatric disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.